CLINICAL TRIAL: NCT00323661
Title: COGNITION - Cognitive Performance & Closed Loop Stimulation
Brief Title: Closed Loop Stimulation, Cognitive Performance, and Quality of Life in Pacemaker Patients
Acronym: COGNITION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BA079
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Cardiac Pacing, Artificial
Keywords: Pacing; Rate-adaptive; Quality of life; Cognitive performance; Atrial fibrillation; Pacemaker sensor
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): Rate-adaptation by Closed Loop Stimulation
  Interventions: Device: Rate-adaptive pacemaker: Closed Loop Stimulation
- 2 (Active Comparator): Accelerometer based pacing rate adaptation
  Interventions: Device: Rate-adaptive pacemaker: accelerometer

INTERVENTIONS:
Device: Rate-adaptive pacemaker: accelerometer — Accelerometer based pacing rate adaptation
  Arms: 2
Device: Rate-adaptive pacemaker: Closed Loop Stimulation — Closed Loop Stimulation (CLS) is a unique concept in rate-adaptive pacing that uses the natural cardiovascular control loop to determine the appropriate pacing rate. Closed Loop Stimulation is the only rate-adaptive system responding to mental stress and thereby assuring optimal cerebral perfusion in everyday activity.
  Arms: 1

SUMMARY:
The purpose of this study is to compare the influence of accelerometer-based rate adaptation and Closed Loop Stimulation on cognitive performance and quality of life in pacemaker patients.

DETAILED DESCRIPTION:
Within the scope of a usual follow-up schedule the influence of the mode of rate-adaptation on cognitive performance of pacemaker patients will be analysed. Accelerometer sensor will be compared with Closed Loop Stimulation over 2 years. The cognitive performance will be measured by means of a standardized psychometric test. The occurrence of atrial fibrillation and serious adverse events, patient self-assessment and quality of life will be evaluated. An analysis of the telemonitored (Home Monitoring) data will be performed in order to identify predictors of changes or differences in cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a CYLOS pacemaker (implantation within the last 3 to 6 weeks)
* Closed Loop Stimulation mode activated since pre-hospital discharge
* Patients with chronotropic incompetence according to physician's judgment
* Maximum sinus rate < 100 beats per minute (bpm) OR percentage of atrial pacing ≥ 25%
* Patients suitable for rate-adaptive pacing for at least 2 years
* Patient informed consent

Exclusion Criteria:

* Age under 55
* Pregnant and breast-feeding women
* Patients who are already enrolled in another study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2006-05; Primary Completion 2010-11 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Cognitive performance assessed by the Number Connection Test | 24 months

SECONDARY OUTCOMES:
Quality of life assessed by the SF-08 | 12 months and 24 months
occurrence of atrial fibrillation | 12 months and 24 months
occurrence of serious adverse events | 12 months and 24 months
self-assessment of general well-being, mental and physical performance assessed by Visual Analogue Scales | 12 months and 24 months
Home Monitoring data | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Wiegand, Prof. Dr., Principal Investigator — Sana-Klinikum Remscheid, 42859 Remscheid, Germany
Locations (55):
- Sydney Adventist Hospital, Sydney, Australia
- Austria (4):
  - A.ö. Krankenhaus der Stadt Linz, Linz
  - Krankenhaus der Barmherzigen Schwestern Ried, Ried
  - A. ö. Landeskrankenhaus Steyr, Steyr
  - Wilhelminenspital der Stadt Wien, Vienna
- Brazil (3):
  - Hospital Anchieta, Instituto do Coracao de Taguatinga, Brasilia - DF
  - Hospital Sao Francisco, Porto Alegre
  - Hospital Real e Benemerita Sociedade Portuguesa de Beneficencia, São Paulo
- Canada (5):
  - Practice Dr. Bloomberg, Burnaby, B.C.
  - Kelowna Cardiology Research, Kelowna BC
  - Hopital Sacre-Coeur, Montreal
  - Dr. Dante Manyauri, Surrey BC
  - Scarborough Cardiology Research, Toronto, Ontario
- Fakultni Nemocnice u Svety Anny, Brno, Czechia
- Germany (35):
  - Universitätsklinik der RWTH Aachen, Aachen
  - Städtische Kliniken Bielefeld, Klinikum Mitte, Bielefeld
  - St. Agnes Hospital GmbH, 1. Medizinische Klinik-Kardiologie, Bocholt
  - Klinikum Coburg, Coburg
  - Klinikum Lippe-Detmold, Detmold
  - Med. Klinik/Kardiologie, Herzzentrum, Universitätsklinik an der Technischen Universität Dresden, Dresden
  - Kreisklinik Ebersberg GmbH, Ebersberg
  - Marien-Hospital Erftstadt-Frauenthal, Erftstadt-Frauenthal
  - Klinken Erlabrunn GmbH, Erlabrunn
  - Westdeutsches Herzzentrum Essen; Klinik für Kardiologie und Thorax-Kardiovaskuläre Chirurgie des Universitätsklinikums Essen, Essen
  - Kardiologisches Zentrum am Zoo, Frankfurt
  - St. Elisabeth-Hospital, Gütersloh
  - Klinikum der Medizinischen Fakultät Halle-Wittenberg, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Zentrum für Kardiologische und Angiologische Medizin Hamburg, Hamburg
  - AK Altona, Hamburg
  - St. Vinzenz-Krankenhaus Hanau gGmbH, Hanau
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum Herford, Herford
  - Evangelisches Krankenhaus Holzminden, Holzminden
  - Klinikum der Universität Jena Klinik für Innere Medizin I, Jena
  - Kardiologische Gemeinschaftspraxis, Kiel
  - Städtisches Klinikum St. Georg, Leipzig
  - Universitätsklinikum Lübeck, Lübeck
  - Krankenhaus St. Franziskus, Medizinische Klinik II, Mönchengladbach
  - St. Vincenz-Krankenhaus GmbH, Paderborn
  - Kardiologische Praxis, Papenburg
  - Christl. Krankenhaus Quakenbrück, Quakenbrück
  - Elisabeth Krankenhaus GmbH, Recklinghausen
  - St. Adolf-Stift, Reinbek
  - Gemeinschaftspraxis Dr. Stenzel/Dr. Ebert, Riesa
  - Evangelisches Elisabeth Krankenhaus, Trier
  - Gemeinschaftspraxis Drs. Schley, Burkhard-Meier, Schemeitat, Viersen
  - Universitätsklinikum Würzburg, Würzburg
- Hong Kong (2):
  - Princess Margaret Hospital, Hong Kong
  - Yan Chai Hospital, Hong Kong
- Wolfson Medical Center, Holon, Israel
- Slovakia (2):
  - Nemocnica Ministerstva Obrany, Bratislava
  - VUSCH East Slovak Cardiology Institute, Arytmology, Košice
- Hospital Universitario La Fé, Valencia, Spain

REFERENCES:
- [Background] Wiegand U, Nuernberg M, Maier SK, Weiss C, Sancho-Tello MJ, Hartmann A, Schuchert A, Maier P, Chan NY. The COGNITION study rationale and design: influence of closed loop stimulation on cognitive performance in pacemaker patients. Pacing Clin Electrophysiol. 2008 Jun;31(6):709-13. doi: 10.1111/j.1540-8159.2008.01075.x. PMID 18507543